CLINICAL TRIAL: NCT00896181
Title: A Phase 2 Study of Sequential and Concurrent Chemoradiation for Patients With Advanced Nasopharyngeal Carcinoma (NPC)
Brief Title: Phase 2 Sequential and Concurrent Chemoradiation for Advanced Nasopharyngeal Carcinoma (NPC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, A. Dimitrios Colevas, Professor of Medicine (Oncology), Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-15411; NCI-2009-01162 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000671087; 8209 (Other: CTEP); ENT0025 (Other: OnCore); NCT00841997 (obsolete NCT alias)
Record Dates: First submitted 2009-05-07; First posted 2009-05-11 (Estimated); Results first posted 2021-04-06 (Actual); Last update posted 2021-04-06 (Actual); Status verified 2021-03

CONDITIONS: Stage II Lymphoepithelioma of the Nasopharynx; Stage II Squamous Cell Carcinoma of the Nasopharynx; Stage III Lymphoepithelioma of the Nasopharynx; Stage III Squamous Cell Carcinoma of the Nasopharynx; Stage IV Lymphoepithelioma of the Nasopharynx; Stage IV Squamous Cell Carcinoma of the Nasopharynx
MeSH Terms: interventions — Docetaxel; Cisplatin; Carboplatin; Fluorouracil; Radiotherapy, Conformal; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Chemoradiation for Nasopharyngeal Carcinoma (Experimental): INDUCTION THERAPY: Patients receive docetaxel intravenously (IV) over 60 minutes on Day 1; cisplatin IV over 1 to 3 hours (or carboplatin IV over 30 minutes) on Day 1; and fluorouracil IV continuously over 24 hours on Days 1 to 5. Each cycle is 21 days, with treatment consisting of up to 3 cycles in the absence of disease progression or unacceptable toxicity.
  CONCURRENT CHEMO-RADIOTHERAPY: Beginning within 3 to 6 weeks after initiating the last course of induction chemotherapy, patients undergo 3-dimensional conformal or intensity-modulated radiotherapy once daily for 6.5 to 7 weeks. Patients also receive cisplatin IV over 1 hour (or carboplatin IV over 30 minutes) once weekly in weeks 1 to 6 in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: docetaxel; Drug: cisplatin; Drug: carboplatin; Drug: fluorouracil; Radiation: 3-dimensional conformal radiation therapy; Radiation: intensity-modulated radiation therapy

INTERVENTIONS:
Drug: docetaxel — Given IV
  Other Names: RP 56976; Taxotere; TXT
Drug: cisplatin — Given IV
  Other Names: CACP; CDDP; CPDD; DDP
Drug: carboplatin — Given IV
  Other Names: Carboplat; CBDCA; JM-8; Paraplat; Paraplatin
Drug: fluorouracil — Given IV
  Other Names: 5-fluorouracil; 5-Fluracil; 5-FU
Radiation: 3-dimensional conformal radiation therapy — Undergo 3-dimensional conformal or intensity-modulated radiotherapy
  Other Names: 3D conformal radiation therapy; 3D-CRT
Radiation: intensity-modulated radiation therapy — Undergo 3-dimensional conformal or intensity-modulated radiotherapy
  Other Names: IMRT

SUMMARY:
This phase 2 trial is studying whether giving a combination of docetaxel, cisplatin, and fluorouracil chemotherapy followed by the combination of cisplatin with radiation therapy works in treating patients with advanced nasopharyngeal cancer. Drugs used in chemotherapy, such as docetaxel, cisplatin, and fluorouracil, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill tumor cells. Specialized radiation therapy that delivers a high dose of radiation directly to the tumor may kill more tumor cells and cause less damage to normal tissue. Giving combination chemotherapy together with radiation therapy may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

• To establish the progression free survival rate at 2 years, using RECIST criteria, to induction treatment with docetaxel, cisplatin, and fluorouracil (TPF) followed by chemoradiotherapy of locoregionally advanced nasopharyngeal carcinoma (NPC)

SECONDARY OBJECTIVE:

• To evaluate complete response rates, safety and feasibility of TPF followed by chemoradiation in patients with NPC

OUTLINE: This is a single site study.

INDUCTION THERAPY: Patients receive docetaxel intravenously (IV) over 60 minutes on Day 1; cisplatin IV over 1 to 3 hours (or carboplatin IV over 30 minutes) on Day 1; and fluorouracil IV continuously over 24 hours on Days 1 to 5. Each cycle is 21 days, with treatment consisting of up to 3 cycles in the absence of disease progression or unacceptable toxicity.

CONCURRENT CHEMO-RADIOTHERAPY: Beginning within 3 to 6 weeks after initiating the last course of induction chemotherapy, patients undergo 3-dimensional conformal or intensity-modulated radiotherapy once daily for 6.5 to 7 weeks. Patients also receive cisplatin IV over 1 hour (or carboplatin IV over 30 minutes) once weekly in weeks 1 to 6 in the absence of disease progression or unacceptable toxicity.

All study treatment is admininstered over the course of 21 weeks. After completion of study treatment, patients are followed periodically for 24 months.

ELIGIBILITY:
INCLUSION CRITERIA

* Histologically- or cytologically-confirmed nasopharyngeal carcinoma meeting the following criteria:

  * WHO type I, II, or III
  * Stage II to IVB disease (minimally T2a, N0, M0 or any T any, N1, M0)
  * Measurable disease, defined as ≥ 1 lesion that can be accurately measured in ≥ 1 dimension as ≥ 20 mm by conventional techniques or as ≥ 10 mm by spiral CT scan
  * Prior diagnostic surgery(s) at the primary site or neck allowed provided there is still measurable disease present
  * Without known brain metastases
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 1
* Life expectancy > 3 months
* Absolute neutrophil count (ANC) ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Total bilirubin ≤ 1.5 times upper limit of normal (ULN)
* Aspartate aminotransferase (AST) / alanine aminotransferase (ALT) ≤ 2.5 times ULN
* Creatinine ≤ 1.5 mg/dL or creatinine clearance ≥ 55 mL/min (NOTE: * Patients with creatinine > grade 1 but < grade 3, hearing loss ≥ grade 2, and peripheral neuropathy ≥ grade 2 are eligible provided they receive carboplatin in place of cisplatin throughout study treatment)
* Hearing loss < grade 2. Hearing loss grade 2 or greater attributable to tumor obstruction, when the bone conduction in the audiogram is consistent with less than grade 2, is permissible for cisplatin. Hearing loss will be evaluated by hearing in the best ear. If hearing loss is grade 2, patients are still eligible but should receive carboplatin throughout the protocol instead of cisplatin.
* Peripheral motor/sensory neuropathy < grade 2. If peripheral neuropathy is grade 2, patients are still eligible but should receive carboplatin throughout the protocol instead of cisplatin.
* Fertile patients must use effective contraception prior to and during study treatment

EXCLUSION CRITERIA

* Uncontrolled intercurrent illness including, but not limited to, any of the following:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Psychiatric illness or social situations that preclude compliance with study requirements
  * Clinically-significant cardiovascular disease
  * Cerebrovascular accident within the past 6 months
  * Myocardial infarction or unstable angina within the past 6 months
  * New York Heart Association (NYHA) class II to IV congestive heart failure
  * Serious and inadequately controlled cardiac arrhythmia
  * Significant vascular disease (eg, aortic aneurysm, history of aortic dissection)
  * Clinically-significant peripheral vascular disease
* History of allergic reaction attributed to compounds of similar chemical or biologic composition to docetaxel, cisplatin, carboplatin, fluorouracil, bevacizumab, or other agents used in this study
* Known brain metastases
* Concurrent combination antiretroviral therapy for HIV-positive patients
* Prior chemotherapy or radiotherapy for nasopharyngeal carcinoma
* Pregnant or nursing

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2008-12-10 (Actual); Primary Completion 2020-01-03 (Actual); Study Completion 2020-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Colevas, Principal Investigator — Stanford University Hospitals and Clinics
Locations (1):
- Stanford University Hospitals and Clinics, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jun M, Pinto H, Le QT, Quon A, Hara W, Coty J, McMillan A, Lu R, Winters E, Lira R, Colevas AD. In search for optimal induction chemotherapy for advanced nasopharyngeal cancer: Standard dosing of Docetaxel, Platinum, and 5-Fluorouracil (TPF) followed by chemoradiation. PLoS One. 2023 Feb 2;18(2):e0276651. doi: 10.1371/journal.pone.0276651. eCollection 2023. PMID 36730145

RESULTS

PARTICIPANT FLOW:
Groups:
- Chemoradiation for Nasopharyngeal Carcinoma: Induction therapy as described, consisting of docetaxel, cisplatin, and fluorouracil Concurrent chemo-radiotherapy as described, 3-dimensional radiotherapy once daily for 6.5 to 7 weeks, with cisplatin weekly.
  The total treatment course is up to 21 weeks.
Period: Overall Study
Arm/Group | Chemoradiation for Nasopharyngeal Carcinoma
Started | 26
Completed | 26
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Chemoradiation for Nasopharyngeal Carcinoma
Number analyzed (Participants) | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 22
  >=65 years | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.3 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 26
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 21
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 26

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Progression-free Survival (PFS) at 2 Years After Chemo-radiotherapy
Description: Progression-free survival (PFS) means to remain alive without disease progression. Progression is defined as either the appearance of one or more new cancer lesions, or a ≥ 20% increase in the sum of the longest diameters (LD) of target cancer lesions, compared the same measurement obtained at the start of treatment. This outcome reported as the number of patients remaining alive at 2 years following chemo-radiotherapy without disease progression, a number without dispersion.
Time Frame: up to 29 months (ie, 24 months post-chemoradiation)
Population: The outcome results are reported by baseline strata, ie, M0 (non-metastatic lesions) and M1 (metastatic lesions).
Measure: Count of Participants; unit: Participants
Arm/Group | Chemoradiation for Nasopharyngeal Carcinoma
Number analyzed (Participants) | 26
Participants
  M0 (non-metastatic lesion): number analyzed (Participants) | 20
  M0 (non-metastatic lesion) | 18
  M1 (metastatic lesion): number analyzed (Participants) | 6
  M1 (metastatic lesion) | 4

2. Primary Outcome: Median Progression-free Survival (PFS)
Description: Progression-free survival (PFS) means to remain alive without disease progression. Progression is defined as either the appearance of one or more new cancer lesions, or a ≥ 20% increase in the sum of the longest diameters (LD) of target cancer lesions, compared the same measurement obtained at the start of treatment. This outcome reported as the median duration of PFS in months since chemo-radiotherapy, with full range.
Time Frame: up to 127 months (includes treatment period of up to 5 months)
Population: The outcome results are reported by baseline strata, ie, M0 (non-metastatic lesions) and M1 (metastatic lesions).
Measure: Median (Full Range); unit: months
Arm/Group | Chemoradiation for Nasopharyngeal Carcinoma
Number analyzed (Participants) | 26
months
  M0 (non-metastatic lesion): number analyzed (Participants) | 20
  M0 (non-metastatic lesion) | 76 [15 to 122]
  M1 (metastatic lesion): number analyzed (Participants) | 6
  M1 (metastatic lesion) | 33 [12 to 90]

3. Secondary Outcome: Overall Survival (OS)
Description: Overall survival (OS) was assessed as the duration of time that study participants remained alive after chemoradiotherapy. The outcome is reported as median OS (with full range).
Time Frame: up to 127 months (includes treatment period of up to 5 months)
Population: The outcome results are reported by baseline strata, ie, M0 (non-metastatic lesions) and M1 (metastatic lesions). The per-protocol duration of treatment on study was 5 months, and the outcome is reported as OS (with full range) from that time.
Measure: Median (Full Range); unit: months
Arm/Group | Chemoradiation for Nasopharyngeal Carcinoma
Number analyzed (Participants) | 26
months
  M0 (non-metastatic lesion): number analyzed (Participants) | 20
  M0 (non-metastatic lesion) | 79 [26 to 122]
  M1 (metastatic lesion): number analyzed (Participants) | 6
  M1 (metastatic lesion) | 76 [18 to 101]

4. Secondary Outcome: Number of Participants With Adverse Events Resulting in Treatment Discontinuation
Description: Adverse events during treatment were assessed as whether they were definitely-, probably-, or possibly-related to protocol treatment (ie, adverse reaction). The outcome is reported as the number of participants who discontinued treatment due to an adverse reaction.
Time Frame: 8 months
Measure: Count of Participants; unit: Participants
Arm/Group | Chemoradiation for Nasopharyngeal Carcinoma
Number analyzed (Participants) | 26
Participants | 1

5. Secondary Outcome: Number of Participants With Treatment Response
Description: Participants who completed 1 cycle of docetaxel, cisplatin, and 5-fluorouracil (TPF) were evaluated for response. Response was assessed for lesions designated as target (TL) and non-target (NTL) as complete response (CR), partial response (PR), stable disease (SD), or progressive disease (PD). The outcome is reported as a number without dispersion.
  TL Criterion:
  * CR: Disappearance of lesions
  * PR: 30% decrease in the sum of the longest diameter (LD) of lesions
  * PD: 20% increase in the sum of the LD of lesions, or any new lesion
  * SD: Neither sufficient shrinkage for PR nor sufficient increase for PD
  NTL Criterion:
  * CR: Disappearance of lesions and normalization of tumor marker level
  * PR / SD: Persistence of one or more lesion(s) and/or maintenance of tumor marker level above the normal limits (includes "incomplete response / PR).
  * PD: Appearance of one or more new lesions and/or unequivocal progression of existing lesions.
Time Frame: up to 29 months (ie, 24 months post-chemoradiation)
Population: The outcome results are reported by baseline strata, ie, M0 (non-metastatic lesions) and M1 (metastatic lesions).
Measure: Count of Participants; unit: Participants
Arm/Group | Chemoradiation for Nasopharyngeal Carcinoma
Number analyzed (Participants) | 26
Participants
  CR for M0 (non-metastatic lesion): number analyzed (Participants) | 20
  CR for M0 (non-metastatic lesion) | 17
  PR for M0 (non-metastatic lesion): number analyzed (Participants) | 20
  PR for M0 (non-metastatic lesion) | 3
  SD for M0 (non-metastatic lesion): number analyzed (Participants) | 20
  SD for M0 (non-metastatic lesion) | 0
  PD for M0 (non-metastatic lesion): number analyzed (Participants) | 20
  PD for M0 (non-metastatic lesion) | 0
  CR for M1 (metastatic lesion): number analyzed (Participants) | 6
  CR for M1 (metastatic lesion) | 3
  PR for M1 (metastatic lesion): number analyzed (Participants) | 6
  PR for M1 (metastatic lesion) | 1
  SD for M1 (metastatic lesion): number analyzed (Participants) | 6
  SD for M1 (metastatic lesion) | 0
  PD for M1 (metastatic lesion): number analyzed (Participants) | 6
  PD for M1 (metastatic lesion) | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected for up to 104 months and All-Cause Mortality was collected up to 127 months.
Arm/Group | Chemoradiation for Nasopharyngeal Carcinoma
All-Cause Mortality (participants affected / at risk) | 4/26
Serious Adverse Events (participants affected / at risk) | 5/26
Other Adverse Events (participants affected / at risk) | 24/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chemoradiation for Nasopharyngeal Carcinoma (N=26)
Febrile Neutropenia (Blood and lymphatic system disorders) | 5 (6)
Gastric Hemorrhage (Blood and lymphatic system disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Thrombocytopenia (Investigations) | 1 (2)
Fatigue (asthenia) (General disorders) | 1 (1)
Thromboemobolic event (Vascular disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chemoradiation for Nasopharyngeal Carcinoma (N=26)
Neuropathy (Nervous system disorders) | 2 (6)
Hearing Impaired (Ear and labyrinth disorders) | 2 (26)
Neutropenia (Blood and lymphatic system disorders) | 12 (22)
Platelet Count Decreased (Investigations) | 7 (12)
Anemia (Blood and lymphatic system disorders) | 11 (56)
Oral Mucositis (Gastrointestinal disorders) | 24 (96)
Abdominal Distension (Gastrointestinal disorders) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
Acid Reflux (Gastrointestinal disorders) | 1 (1)
Alanine Aminotransferace Increase (Investigations) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 4 (15)
Anorexia (Metabolism and nutrition disorders) | 4 (13)
Constipation (Gastrointestinal disorders) | 1 (1)
Infections and infestations - Other, Coronavirus (Infections and infestations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 4 (4)
Dermatitis (Skin and subcutaneous tissue disorders) | 11 (18)
Dermatitis radiation (Injury, poisoning and procedural complications) | 5 (7)
Diarrhea (Gastrointestinal disorders) | 4 (4)
Dysgeusia (Nervous system disorders) | 6 (32)
Dysphagia (Gastrointestinal disorders) | 7 (15)
Fatigue (General disorders) | 10 (27)
Febrile Neutropenia (Blood and lymphatic system disorders) | 4 (5)
Hyperglycemia (Metabolism and nutrition disorders) | 5 (14)
Hypoalbuminemia (Metabolism and nutrition disorders) | 5 (12)
Hypocalcemia (Metabolism and nutrition disorders) | 3 (8)
Hypokalemia (Metabolism and nutrition disorders) | 2 (4)
Lymphocyte count decreased (Investigations) | 18 (114)
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 8 (18)
Oral Pain (Gastrointestinal disorders) | 4 (16)
Pain in Extremities (Musculoskeletal and connective tissue disorders) | 1 (1)
Palmar Plantar Syndrome (Skin and subcutaneous tissue disorders) | 1 (2)
Paresthesia (Nervous system disorders) | 1 (12)
Salivary Duct Inflammation (Gastrointestinal disorders) | 2 (2)
Skin Infection (Infections and infestations) | 1 (2)
Somnolence (Nervous system disorders) | 1 (1)
Infections and infestations - Other, Thrush (Infections and infestations) | 1 (1)
Typhlitis (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3)
Weight Loss (Investigations) | 7 (18)
White blood cell count decreased (Investigations) | 8 (16)
Xerostomia (Gastrointestinal disorders) | 4 (16)
Neutropenia (Blood and lymphatic system disorders) | 3 (7)
Creatinine Increased (Investigations) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Otitis Media (Infections and infestations) | 1 (1)
Otitis Externa (Infections and infestations) | 1 (1)
Salivary Duct Inflammation (Gastrointestinal disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, skin changes (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, skin problems (Skin and subcutaneous tissue disorders) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Laryngeal Inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypertension (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-12-05): https://cdn.clinicaltrials.gov/large-docs/81/NCT00896181/Prot_SAP_000.pdf